CLINICAL TRIAL: NCT02132494
Title: Active Smarter Kids: A Cluster-randomized Controlled Trial Investigating the Effect of Daily Physical Activity on Children's Academic Performance and on Risk Factors for Lifestyle-related Non-communicable Diseases
Brief Title: Active Smarter Kids: A Cluster-randomized Controlled Trial
Acronym: ASK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Western Norway University of Applied Sciences (Other)
Collaborators: The Research Council of Norway (Other)
Responsible Party: Principal Investigator, Eivind Aadland, Associate professor, Western Norway University of Applied Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HISF_2014; 2013/1893 (Registry Identifier: The South-East A Regional Committees for Medical and Health Research Ethics (Norway))
Record Dates: First submitted 2014-04-07; First posted 2014-05-07 (Estimated); Last update posted 2019-10-02 (Actual); Status verified 2019-10

CONDITIONS: Academic Performance; Primary Prevention; Physical Activity
MeSH Terms: conditions — Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Physical activity (Experimental): 60 minutes of daily physical activity during one school year
  Interventions: Behavioral: Physical activity
- Control (No Intervention)

INTERVENTIONS:
Behavioral: Physical activity
  Arms: Physical activity

SUMMARY:
The relationship between physical activity and academic performance has received widespread attention owing to the pressure on schools to graduate pupils who meet accepted academic standards. As important, there are global concerns regarding the increased prevalence of lifestyle-related non-communicable diseases (NCDs). First, Norway has a history of mediocre scores on international comparative academic performance tests such as Trends in International Mathematics and Science Study (TIMSS) and the Programme for International Student Assessment (PISA) [1]. It is therefore important to develop and evaluate strategic programs that may enhance pupil's academic performance. It is increasingly evident that a physical activity strategy that brings about enhanced cognitive function, better blood flow, and more, plays a key role in this effort [2]. Second, the prevalence of NCDs, such as diabetes mellitus type 2, is increasing worldwide, and such NCDs affect people of all ages [3]. Hence, healthcare costs are escalating to unaffordable levels. The best means to deal with this immense problem is through primary prevention, and physical activity is a powerful common denominator known to play a key role in preventing a host of NCDs [4].

Consequently, both World Health Organization (WHO) and the Norwegian health authorities call for effective primary prevention strategies to promote physical activity in children and adolescents [5, 6]. Prop. 90 L (2010-2011) Act on public health work [6] emphasizes that physical activity in school can benefit both the learning process and public health prevention.

Therefore, the objective of the ASK-study is to investigate the effects on academic performance of 60 minutes of daily physical activity during one school year. Furthermore, due to the complexity in the relationship between physical activity and academic performance, it is necessary to identify possible mediating and moderating variables as cognitive performance, quality of life (QoL), classroom behavior, motor skills and motivation. Also, we aim to investigate changes in risk factors related to NCDs and factors that influence NSDs, such as physical activity, sedentary behavior and health-related fitness.

In addition a qualitative part of the ASK-Study will be conducted to get an in-depth understanding of the children's embodied experiences and the meaning of the social learning culture in school physical activity (PA). This will give us an in-depth description of the intervention context, offer insight in how the intervention possibly influences children's overall development and enables us to estimate potential long term effects of the intervention.

If successful, the ASK cluster-randomized controlled trial (RCT) could provide much needed solutions to enhancing schoolchildren's academic performance and position the school as an effective setting for a massive public health intervention concerning the prevention of NCDs.

ELIGIBILITY:
Inclusion Criteria:

* all children attending 5th grade at the invited schools in Sogn og Fjordane county (Norway) during the school-year 2014/2015

Exclusion Criteria:

* those children whom for language barriers are unable to perform national tests in Numeracy, Norwegian and English

Ages: 8 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1202 (Actual)
Dates: Start 2014-03; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Academic performance | October 2014 - June 2015 (8 months)
  Academic performance will be measured by Norwegian "national tests" in Numeracy, Norwegian and English

SECONDARY OUTCOMES:
Risk factors for lifestyle-related non-communicable diseases (NCDs) | August 2014 - June 2015 (10 months)
  We will measure physical activity, sedentary behavior, health-related physical fitness, measures of adiposity, blood pressure and biomarkers for metabolic health
Executive functions | August 2014 - June 2015 (10 months)
  Inhibition, working memory and cognitive flexibility will be assessed by pen-and-paper testing
Qualitative study of embodied experiences and interpersonal relations | August 2014 - June 2015 (10 months)
  Qualitative methods will be used to explore how children act in the context of physical education and the ASK-intervention, and how their experiences are constructed in the interaction between individual and social factors. We will also explore to what extent children are capable to reflect over their bodily and social experiences.

OTHER OUTCOMES:
Quality of life and well-being | August 2014 - June 2015 (10 months)
  We will measure self-reported physical well-being, psychological well-being, autonomy & parent relation, social support & peers and school environment.

CONTACTS AND LOCATIONS:
Overall Officials: Sigmund A Anderssen, PhD, Principal Investigator — Sogn og Fjordande University College
Locations (1):
- Sogn og Fjordane University College, Sogndal, Sogn Og Fjordane, Norway

REFERENCES:
- [Background] 1. Kjærnsli, M., Tid for tunge løft: norske elevers kompetanse i naturfag, lesing og matematikk i PISA 2006. 2007, Oslo: Universitetsforl.
- [Background] Singh A, Uijtdewilligen L, Twisk JW, van Mechelen W, Chinapaw MJ. Physical activity and performance at school: a systematic review of the literature including a methodological quality assessment. Arch Pediatr Adolesc Med. 2012 Jan;166(1):49-55. doi: 10.1001/archpediatrics.2011.716. PMID 22213750
- [Background] 3. WHO, World Health Organization. Prevention and control of noncommunicable diseases: implementation of the global strategy. 2008, WHO: Geneva.
- [Background] 4. WHO, World Health Organization [cited 2013 15.08]; Available from: http://www.euro.who.int/en/what-we-do/health-topics/disease-prevention/physical-activity/facts-and-figures/10-key-facts-on-physical-activity-in-the-who-european-region. 2011, WHO.
- [Background] 5. WHO, World Health Organization. Global Strategy on Diet, Physical Activity and Health. 57th World Health Assembly. 2004, WHO: Geneva.
- [Background] 6. PttSL, (2010-2011) Act on public health work.Lov om Folkehelsearbeid. 2010
- [Derived] Jones PR, Rajalahti T, Resaland GK, Aadland E, Steene-Johannessen J, Anderssen SA, Bathen TF, Andreassen T, Kvalheim OM, Ekelund U. Associations of lipoprotein particle profile and objectively measured physical activity and sedentary time in schoolchildren: a prospective cohort study. Int J Behav Nutr Phys Act. 2022 Jan 21;19(1):5. doi: 10.1186/s12966-022-01244-w. PMID 35062967
- [Derived] Rajalahti T, Aadland E, Resaland GK, Anderssen SA, Kvalheim OM. Influence of adiposity and physical activity on the cardiometabolic association pattern of lipoprotein subclasses to aerobic fitness in prepubertal children. PLoS One. 2021 Nov 18;16(11):e0259901. doi: 10.1371/journal.pone.0259901. eCollection 2021. PMID 34793516
- [Derived] Stavnsbo M, Aadland E, Anderssen SA, Chinapaw M, Steene-Johannessen J, Andersen LB, Resaland GK. Effects of the Active Smarter Kids (ASK) physical activity intervention on cardiometabolic risk factors in children: A cluster-randomized controlled trial. Prev Med. 2020 Jan;130:105868. doi: 10.1016/j.ypmed.2019.105868. Epub 2019 Oct 22. PMID 31654725
- [Derived] Aadland E, Kvalheim OM, Anderssen SA, Resaland GK, Andersen LB. Multicollinear physical activity accelerometry data and associations to cardiometabolic health: challenges, pitfalls, and potential solutions. Int J Behav Nutr Phys Act. 2019 Aug 27;16(1):74. doi: 10.1186/s12966-019-0836-z. PMID 31455305
- [Derived] Aadland E, Kvalheim OM, Anderssen SA, Resaland GK, Andersen LB. The multivariate physical activity signature associated with metabolic health in children. Int J Behav Nutr Phys Act. 2018 Aug 15;15(1):77. doi: 10.1186/s12966-018-0707-z. PMID 30111365
- [Derived] Aadland E, Andersen LB, Ekelund U, Anderssen SA, Resaland GK. Reproducibility of domain-specific physical activity over two seasons in children. BMC Public Health. 2018 Jul 3;18(1):821. doi: 10.1186/s12889-018-5743-8. PMID 29970050
- [Derived] Aadland KN, Aadland E, Andersen JR, Lervag A, Moe VF, Resaland GK, Ommundsen Y. Executive Function, Behavioral Self-Regulation, and School Related Well-Being Did Not Mediate the Effect of School-Based Physical Activity on Academic Performance in Numeracy in 10-Year-Old Children. The Active Smarter Kids (ASK) Study. Front Psychol. 2018 Feb 28;9:245. doi: 10.3389/fpsyg.2018.00245. eCollection 2018. PMID 29541050
- [Derived] Aadland E, Andersen LB, Anderssen SA, Resaland GK. A comparison of 10 accelerometer non-wear time criteria and logbooks in children. BMC Public Health. 2018 Mar 6;18(1):323. doi: 10.1186/s12889-018-5212-4. PMID 29510709
- [Derived] Aadland E, Andersen LB, Skrede T, Ekelund U, Anderssen SA, Resaland GK. Reproducibility of objectively measured physical activity and sedentary time over two seasons in children; Comparing a day-by-day and a week-by-week approach. PLoS One. 2017 Dec 7;12(12):e0189304. doi: 10.1371/journal.pone.0189304. eCollection 2017. PMID 29216318
- [Derived] Resaland GK, Moe VF, Bartholomew JB, Andersen LB, McKay HA, Anderssen SA, Aadland E. Gender-specific effects of physical activity on children's academic performance: The Active Smarter Kids cluster randomized controlled trial. Prev Med. 2018 Jan;106:171-176. doi: 10.1016/j.ypmed.2017.10.034. Epub 2017 Dec 1. PMID 29104022
- [Derived] Aadland KN, Ommundsen Y, Aadland E, Bronnick KS, Lervag A, Resaland GK, Moe VF. Executive Functions Do Not Mediate Prospective Relations between Indices of Physical Activity and Academic Performance: The Active Smarter Kids (ASK) Study. Front Psychol. 2017 Jun 29;8:1088. doi: 10.3389/fpsyg.2017.01088. eCollection 2017. PMID 28706500
- [Derived] Skrede T, Stavnsbo M, Aadland E, Aadland KN, Anderssen SA, Resaland GK, Ekelund U. Moderate-to-vigorous physical activity, but not sedentary time, predicts changes in cardiometabolic risk factors in 10-y-old children: the Active Smarter Kids Study. Am J Clin Nutr. 2017 Jun;105(6):1391-1398. doi: 10.3945/ajcn.116.150540. Epub 2017 Apr 5. PMID 28381476
- [Derived] Resaland GK, Aadland E, Moe VF, Aadland KN, Skrede T, Stavnsbo M, Suominen L, Steene-Johannessen J, Glosvik O, Andersen JR, Kvalheim OM, Engelsrud G, Andersen LB, Holme IM, Ommundsen Y, Kriemler S, van Mechelen W, McKay HA, Ekelund U, Anderssen SA. Effects of physical activity on schoolchildren's academic performance: The Active Smarter Kids (ASK) cluster-randomized controlled trial. Prev Med. 2016 Oct;91:322-328. doi: 10.1016/j.ypmed.2016.09.005. Epub 2016 Sep 7. PMID 27612574
- [Derived] Resaland GK, Moe VF, Aadland E, Steene-Johannessen J, Glosvik O, Andersen JR, Kvalheim OM, McKay HA, Anderssen SA; ASK study group. Active Smarter Kids (ASK): Rationale and design of a cluster-randomized controlled trial investigating the effects of daily physical activity on children's academic performance and risk factors for non-communicable diseases. BMC Public Health. 2015 Jul 28;15:709. doi: 10.1186/s12889-015-2049-y. PMID 26215478